CLINICAL TRIAL: NCT01405521
Title: Understanding Typhoid Disease After Vaccination: a Single Centre, Randomised, Doubleblind, Placebo Controlled Study to Evaluate M01ZH09 in a Healthy Adult Challenge Model, Using Ty21a Vaccine as a Positive Control.
Brief Title: Understanding Typhoid Disease After Vaccination
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Wellcome Trust (Other); Imperial College London (Other); University of Maryland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OVG 2011/02; 2011-000381-35 (EudraCT Number)
Record Dates: First submitted 2011-07-28; First posted 2011-07-29 (Estimated); Last update posted 2023-05-06 (Actual); Status verified 2020-12

CONDITIONS: Typhoid Fever; Enteric Fever; Typhoid
Keywords: typhoid vaccine M01ZH09; Ty21a typhoid vaccine
MeSH Terms: conditions — Typhoid Fever | interventions — Ty21a typhoid vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- M01ZH09 vaccine (Experimental)
  Interventions: Biological: M10ZH09 vaccine
- Vaccine placebo (Placebo Comparator)
  Interventions: Biological: Vaccine placebo (excipients only)
- Ty21a vaccine (Other): Positive control
  Interventions: Biological: Ty21a

INTERVENTIONS:
Biological: Vaccine placebo (excipients only) — single oral dose,
  Arms: Vaccine placebo
Biological: Ty21a — 3 oral doses, alternate days
  Other Names: Vivotif
  Arms: Ty21a vaccine
Biological: M10ZH09 vaccine — single oral dose
  Other Names: Typhella
  Arms: M01ZH09 vaccine

SUMMARY:
Using an established model of human typhoid infection, whereby healthy adults are deliberately infected with typhoid-causing bacteria, the investigators will determine how effective a new oral typhoid vaccine (M01ZH09) is in preventing infection. A previously licensed oral typhoid vaccine (Ty21a) will be used to make sure the challenge model used works properly.

DETAILED DESCRIPTION:
Typhoid is a serious infection killing up to 600,000 people every year; it is a frequent cause of fever and hospital admission in areas where disease is common. As the infection is restricted to humans, it should be possible to eliminate typhoid; better vaccines and ways of confirming infection are required in order for this to succeed. We propose to use a recently established human typhoid challenge model in order to evaluate a novel oral vaccine candidate and to develop new methods for diagnosing typhoid.

Although there are vaccines available to prevent typhoid, they offer little protection to populations where typhoid predominates, especially young children. Currently, the effectiveness of vaccines against typhoid cannot be predicted, as measures of protection against typhoid are unknown. As a result, implementation of vaccine programmes in disease endemic regions currently requires large and expensive trials in each new population, significantly delaying programmatic implementation.

We will use a typhoid challenge model to achieve our goal of accelerating the introduction of more effective vaccines into populations with a high burden of disease. Healthy adults will be vaccinated with either a novel oral typhoid vaccine or vaccine-placebo prior to being infected with the bacteria causing typhoid. This will allow us to measure the effectiveness of the vaccine and to identify components of the immune response important in producing protection against infection.

Current methods for confirming typhoid infection are slow and insensitive, particularly in endemic regions where the cost of laboratory equipment is prohibitive. In this project, we will also explore ways to diagnose typhoid, with the aim of developing tests that are quick, reliable and are be cost-effective in resource-poor settings. This would improve individual patient management, and allow accurate measurement of disease burden, which is vital to improve the efforts of vaccine programmes.

ELIGIBILITY:
Inclusion criteria:

* Male or female aged 18 - 60 years inclusive and in good health.
* Have an abdominal ultrasound scan result documented demonstrating no evidence of gallbladder pathology.
* Willing to allow their general practitioner and/or hospital consultant (if relevant) and the Health Protection Unit to be notified of participation in the study.
* Agree to refrain from blood donation in the future if diagnosed with typhoid fever.
* Be willing to have 24-hour contact with study staff during the four weeks post-challenge.

Exclusion Criteria:

* Have previously received any typhoid vaccine, been resident in a typhoid endemic country for over 6 months, been diagnosed with probable or confirmed typhoid infection or been challenged with Salmonella Typhi or enrolled in a typhoid challenge study.
* Have any known or suspected impairment or alteration of immune function.
* History of significant cardiovascular disease.
* History of significant respiratory disease.
* History of significant endocrine disorder.
* History of significant renal or bladder disease.
* History of biliary tract disease.
* History of significant gastrointestinal disease.
* History of significant neurological disease.
* History of significant metabolic disease.
* History of significant haematological diagnosis.
* History of psychiatric illness requiring hospitalisation, current known or suspected drug or alcohol misuse.
* History of significant infectious disease.
* History of non-benign cancer.
* Presence of any implants or prostheses.
* Hypersensitivity to any component of the vaccine or are hypersensitive to two or more of the following antibiotics: ciprofloxacin, azithromycin, ampicillin, trimethoprim sulfamethoxazole.
* Female participant who is pregnant, lactating or who is unwilling to ensure that they or their partner use effective contraception one month prior to vaccination and continue to do so until two negative stool samples obtained a week apart, a minimum of 1 week after completion of antibiotic treatment have been obtained.
* Current occupation involving: clinical or social work with direct contact with young children (defined as those attending pre-school groups, nursery or aged less than 2 years); highly susceptible patients or persons in whom typhoid infection would have particularly serious consequences (i.e. those who are immunocompromised or debilitated); care work involving the elderly.
* Current occupation as a commercial food handler involving the preparation or serving of unwrapped foods not subjected to further heating.
* Household contact with a young child (defined as above).
* Household/close contact who is immunocompromised.
* Scheduled elective surgery or other procedures requiring general anaesthesia during the vaccine/challenge period, at time of enrolment.
* Participants who have taken part in other research involving an investigational product (IMP) within the 30 days prior to enrolment.
* Have received blood, blood products and/or plasma derivatives including parenteral immunoglobulin preparations in the previous 3 months
* Any other significant disease or disorder which, in the opinion of the investigator, may put the participants at risk because of participation in the study, may influence the result of the study, or affect the participant's ability to participate in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2011-10-07 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2022-05-06 (Actual)

PRIMARY OUTCOMES:
Diagnosis of typhoid fever | 2 weeks after typhoid challenge
  Typhoid fever defined as development of Gram negative bacteraemia after day 5 or temperature over 38C persisting for 12 hours or more.
  Typhoid challenge defined as ingestion of virulent S. Typhi (Quailes strain).

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Pollard, Principal Investigator — Oxford Vaccine Group, Department of Paediatrics, University of Oxford
Locations (1):
- Oxford Vaccine Group, Centre for Clinical Vaccinology and Tropical Medicine, Oxford, United Kingdom

REFERENCES:
- [Background] Gibani MM, Voysey M, Jin C, Jones C, Thomaides-Brears H, Jones E, Baker P, Morgan M, Simmons A, Gordon MA, Cerundolo V, Pitzer VE, Angus B, Levine MM, Darton TC, Pollard AJ. The Impact of Vaccination and Prior Exposure on Stool Shedding of Salmonella Typhi and Salmonella Paratyphi in 6 Controlled Human Infection Studies. Clin Infect Dis. 2019 Apr 8;68(8):1265-1273. doi: 10.1093/cid/ciy670. PMID 30252031
- [Background] Darton TC, Blohmke CJ, Giannoulatou E, Waddington CS, Jones C, Sturges P, Webster C, Drakesmith H, Pollard AJ, Armitage AE. Rapidly Escalating Hepcidin and Associated Serum Iron Starvation Are Features of the Acute Response to Typhoid Infection in Humans. PLoS Negl Trop Dis. 2015 Sep 22;9(9):e0004029. doi: 10.1371/journal.pntd.0004029. eCollection 2015 Sep. PMID 26394303
- [Background] Juel HB, Thomaides-Brears HB, Darton TC, Jones C, Jones E, Shrestha S, Sie R, Eustace A, Galal U, Kurupati P, Van TT, Thieu NTV, Baker S, Blohmke CJ, Pollard AJ. Salmonella Typhi Bactericidal Antibodies Reduce Disease Severity but Do Not Protect against Typhoid Fever in a Controlled Human Infection Model. Front Immunol. 2018 Jan 17;8:1916. doi: 10.3389/fimmu.2017.01916. eCollection 2017. PMID 29387052
- [Background] Blohmke CJ, Hill J, Darton TC, Carvalho-Burger M, Eustace A, Jones C, Schreiber F, Goodier MR, Dougan G, Nakaya HI, Pollard AJ. Induction of Cell Cycle and NK Cell Responses by Live-Attenuated Oral Vaccines against Typhoid Fever. Front Immunol. 2017 Oct 12;8:1276. doi: 10.3389/fimmu.2017.01276. eCollection 2017. PMID 29075261
- [Background] Barton A, Hill J, Bibi S, Chen L, Jones C, Jones E, Camara S, Shrestha S, Jin C, Gibani MM, Dobinson H, Waddington C, Darton TC, Blohmke CJ, Pollard AJ. Genetic Susceptibility to Enteric Fever in Experimentally Challenged Human Volunteers. Infect Immun. 2022 Apr 21;90(4):e0038921. doi: 10.1128/iai.00389-21. Epub 2022 Mar 7. PMID 35254093
- [Background] Darton TC, Baker S, Randall A, Dongol S, Karkey A, Voysey M, Carter MJ, Jones C, Trappl K, Pablo J, Hung C, Teng A, Shandling A, Le T, Walker C, Molina D, Andrews J, Arjyal A, Basnyat B, Pollard AJ, Blohmke CJ. Identification of Novel Serodiagnostic Signatures of Typhoid Fever Using a Salmonella Proteome Array. Front Microbiol. 2017 Sep 19;8:1794. doi: 10.3389/fmicb.2017.01794. eCollection 2017. PMID 28970824
- [Background] Darton TC, Jones C, Dongol S, Voysey M, Blohmke CJ, Shrestha R, Karkey A, Shakya M, Arjyal A, Waddington CS, Gibani M, Carter MJ, Basnyat B, Baker S, Pollard AJ. Assessment and Translation of the Antibody-in-Lymphocyte Supernatant (ALS) Assay to Improve the Diagnosis of Enteric Fever in Two Controlled Human Infection Models and an Endemic Area of Nepal. Front Microbiol. 2017 Oct 23;8:2031. doi: 10.3389/fmicb.2017.02031. eCollection 2017. PMID 29109704
- [Result] Darton TC, Jones C, Blohmke CJ, Waddington CS, Zhou L, Peters A, Haworth K, Sie R, Green CA, Jeppesen CA, Moore M, Thompson BA, John T, Kingsley RA, Yu LM, Voysey M, Hindle Z, Lockhart S, Sztein MB, Dougan G, Angus B, Levine MM, Pollard AJ. Using a Human Challenge Model of Infection to Measure Vaccine Efficacy: A Randomised, Controlled Trial Comparing the Typhoid Vaccines M01ZH09 with Placebo and Ty21a. PLoS Negl Trop Dis. 2016 Aug 17;10(8):e0004926. doi: 10.1371/journal.pntd.0004926. eCollection 2016 Aug. PMID 27533046
- See also: Oxford Vaccine Group homepage — http://www.ovg.ox.ac.uk/
- See also: Blohmke CJ, Hill J, Darton TC, Carvalho-Burger M, Eustace A, Jones C, Schreiber F, Goodier MR, Dougan G, Nakaya HI, Pollard AJ. Induction of Cell Cycle and NK Cell Responses by Live-Attenuated Oral Vaccines against Typhoid Fever. — https://pubmed.ncbi.nlm.nih.gov/29075261/
- See also: The Impact of Vaccination and Prior Exposure on Stool Shedding of Salmonella Typhi and Salmonella Paratyphi in 6 Controlled Human Infection Studies — https://pubmed.ncbi.nlm.nih.gov/30252031/
- See also: Rapidly Escalating Hepcidin and Associated Serum Iron Starvation Are Features of the Acute Response to Typhoid Infection in Humans — https://pubmed.ncbi.nlm.nih.gov/26394303/
- See also: Salmonella Typhi Bactericidal Antibodies Reduce Disease Severity but Do Not Protect against Typhoid Fever in a Controlled Human Infection Model — https://pubmed.ncbi.nlm.nih.gov/29387052/
- See also: Induction of Cell Cycle and NK Cell Responses by Live-Attenuated Oral Vaccines against Typhoid Fever — https://pubmed.ncbi.nlm.nih.gov/29075261/
- See also: Genetic Susceptibility to Enteric Fever in Experimentally Challenged Human Volunteers — https://pubmed.ncbi.nlm.nih.gov/35254093/
- See also: Identification of Novel Serodiagnostic Signatures of Typhoid Fever Using a Salmonella Proteome Array — https://pubmed.ncbi.nlm.nih.gov/28970824/
- See also: Assessment and Translation of the Antibody-in-Lymphocyte Supernatant (ALS) Assay to Improve the Diagnosis of Enteric Fever in Two Controlled Human Infection Models and an Endemic Area of Nepal — https://pubmed.ncbi.nlm.nih.gov/29109704/